CLINICAL TRIAL: NCT05881434
Title: Influence of a Questionnaire on Patients' Emergency Room Expectations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orange Park Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Expectations
Record Dates: First submitted 2022-01-12; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Emergencies; Satisfaction, Patient; Expectations; Physician-Patient Relations
MeSH Terms: conditions — Emergencies; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expectations Questionnaire (Experimental): Provision of expectations questionnaire and associated instructions to patient.
  Interventions: Other: Emergency Department Visit Expectations Questionnaire
- Control (No Intervention): Usual care (no expectations questionnaire or further instruction)

INTERVENTIONS:
Other: Emergency Department Visit Expectations Questionnaire — Patients presented with novel questionnaire designed to illicit patient's self-reported expectations across four domains (overall purpose of visit, medication intervention, imaging intervention and disposition) during check-in when arriving at the emergency department. Patients instructed to present the completed questionnaire to the treating provider.
  Arms: Expectations Questionnaire

SUMMARY:
The goal of this study is to determine whether a novel questionnaire designed to illicit patient's self-reported expectations across four domains (overall purpose of visit, medication intervention, imaging intervention and disposition) improves patient-provider communication as evaluated by an exit survey during an emergency room visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients who arrive through the ED main entrance (non-EMS)
* Patients aged 18 years and older
* Patients who demonstrate decision making capacity
* Patients who willingly consent to participate

Exclusion criteria:

* Patients in distress (physical, emotional, or other) as determined by investigator
* Patients who demonstrate altered mental status or lack of capacity to consent
* Patients who require immediate medical intervention including diagnostic and/or treatment intervention
* Prisoners and patient under involuntary holds

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-10-17 (Actual)

PRIMARY OUTCOMES:
Patient reported provider understanding of patient's visit expectations | After patient discharge instructions given (or for patients being admitted/transferred, after admission/transfer request), up to 15 minutes after either event
  Q: "My ER provider understood my expectations for my ER visit today" with agreement responses on a 5-point Likert scale (strongly disagree to strongly agree)

SECONDARY OUTCOMES:
Patient reported degree to which visit expectations were met | After patient discharge instructions given (or for patients being admitted/transferred, after admission/transfer request), up to 15 minutes after either event
  Q: "My expectations for my ER visit today were met" with agreement responses on a 5-point Likert scale (strongly disagree to strongly agree)
Patient reported provider courtesy | After patient discharge instructions given (or for patients being admitted/transferred, after admission/transfer request), up to 15 minutes after either event
  Q: "Courtesy of your provider" with response options from Very Poor to Very Good
Patient reported provider listening | After patient discharge instructions given (or for patients being admitted/transferred, after admission/transfer request), up to 15 minutes after either event
  Q: "Your provider took the time to listen to you" with response options from Very Poor to Very Good
Patient reported inclusion in treatment decisions | After patient discharge instructions given (or for patients being admitted/transferred, after admission/transfer request), up to 15 minutes after either event
  Q: "Your provider included you in decisions about your treatment" with response options from Very Poor to Very Good

CONTACTS AND LOCATIONS:
Locations (1):
- Orange Park Medical Center, Orange Park, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided